CLINICAL TRIAL: NCT00002493
Title: WHOLE ABDOMINAL RADIOTHERAPY VERSUS CIRCADIAN-TIMED COMBINATION DOXORUBICIN-CISPLATIN CHEMOTHERAPY IN ADVANCED ENDOMETRIAL CARCINOMA -- PHASE III
Brief Title: Radiation Therapy Compared With Combination Chemotherapy in Treating Patients With Advanced Endometrial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: GOG-0122; CDR0000077572
Record Dates: First submitted 1999-11-01; First posted 2004-08-23 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Endometrial Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: stage III endometrial carcinoma; stage IV endometrial carcinoma; endometrial adenocarcinoma; endometrial adenosquamous cell carcinoma; endometrial adenoacanthoma; endometrial papillary serous carcinoma; endometrial clear cell carcinoma; psychosocial effects of cancer and its treatment
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Cisplatin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: doxorubicin hydrochloride
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which treatment regimen is more effective for endometrial cancer.

PURPOSE: Randomized phase III trial to compare radiation therapy with chemotherapy in treating patients who have advanced endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare overall survival, progression-free interval, and patterns of failure of maximally debulked patients with stage III/IV endometrial carcinoma treated with whole-abdominal irradiation vs. doxorubicin/cisplatin. II. Compare the incidence and type of acute and late adverse events observed with these two treatment regimens. III. Compare changes in fatigue, elimination, and neurologic impairment that impact on quality of life in patients treated with these two regimens. IV. Assess the difference in short-term versus long-term impact on quality of life between the two treatment groups. V. Compare quality-of-life outcomes over time between these two treatment groups.

OUTLINE: Randomized study. Arm I: Radiotherapy. Whole-abdominal irradiation using equipment with photon energies ranging from 6 to 25 MV. Arm II: 2-Drug Combination Chemotherapy. Doxorubicin, DOX, NSC-123127; Cisplatin, CDDP, NSC-119875.

PROJECTED ACCRUAL: It is anticipated that 355 patients will be entered over 7.4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Pathological stage III/IV endometrial carcinoma of any histology (including clear cell and serous papillary carcinomas) The following extent of disease eligible: Positive adnexa Tumor invading the serosa Positive pelvic nodes Positive para-aortic nodes Involvement of the bowel mucosa Intra-abdominal metastases Positive pelvic washings Vaginal involvement within the radiotherapy field Hysterectomy and bilateral salpingo-oophorectomy (BSO) required with residual tumor not greater than 2 cm at any site Selective pelvic and para-aortic lymph node sampling optional for patients with stage III/IV disease by other criteria If para-aortic nodes are positive, scalene nodes must be negative on biopsy and chest CT must be negative for intrathoracic disease The following disease conditions exclude: Parenchymal liver metastasis Lung metastasis Positive inguinal nodes Positive scalene nodes Recurrent disease Protocol therapy must begin within 8 weeks after surgery

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-3 Hematopoietic: WBC at least 3,000/mm3 Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal AST no greater than 3 times normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: Left ventricular ejection fraction normal Other: No past or concomitant malignancy other than nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior chemotherapy Endocrine therapy: Prior progestational agents allowed No other prior endocrine therapy Radiotherapy: No prior pelvic or abdominal radiotherapy Surgery: Hysterectomy and BSO required Pelvic and para-aortic lymph node sampling optional (see Disease Characteristics)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-05; Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus E. Randall, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (58):
- United States (58):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Brookview Research, Inc., Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington

REFERENCES:
- [Background] Moore KN, Tian C, McMeekin DS, Thigpen JT, Randall ME, Gallion HH. Does the progression-free interval after primary chemotherapy predict survival after salvage chemotherapy in advanced and recurrent endometrial cancer?: a Gynecologic Oncology Group ancillary data analysis. Cancer. 2010 Dec 1;116(23):5407-14. doi: 10.1002/cncr.25480. Epub 2010 Aug 24. PMID 20737572
- [Background] Diavolitsis V, Boyle J, Singh DK, Small W Jr. The role of adjuvant radiation in endometrial cancer. Oncology (Williston Park). 2009 Apr 15;23(4):342-9. PMID 19476264
- [Background] Modesitt SC, Tian C, Kryscio R, Thigpen JT, Randall ME, Gallion HH, Fleming GF; Gynecologic Oncology Group. Impact of body mass index on treatment outcomes in endometrial cancer patients receiving doxorubicin and cisplatin: a Gynecologic Oncology Group study. Gynecol Oncol. 2007 Apr;105(1):59-65. doi: 10.1016/j.ygyno.2006.10.045. Epub 2006 Dec 5. PMID 17150247
- [Background] Modesitt S, Tian C, Kryscio R, et al.: Impact of body mass index (BMI) on treatment outcomes in advanced or recurrent endometrial cancer patients receiving doxorubicin/cisplatin chemotherapy: a Gynecologic Oncology Group study. [Abstract] Society of Gynecologic Oncologists, 2006 Annual Meeting on Women's Cancer, March 22-26, 2006, Palm Springs, CA. A-93, 2006.
- [Result] Tewari KS, Filiaci VL, Spirtos NM, Mannel RS, Thigpen JT, Cibull ML, Monk BJ, Randall ME. Association of number of positive nodes and cervical stroma invasion with outcome of advanced endometrial cancer treated with chemotherapy or whole abdominal irradiation: a Gynecologic Oncology Group study. Gynecol Oncol. 2012 Apr;125(1):87-93. doi: 10.1016/j.ygyno.2011.12.414. Epub 2011 Dec 8. PMID 22155678
- [Result] Bruner DW, Barsevick A, Tian C, Randall M, Mannel R, Cohn DE, Sorosky J, Spirtos NM. Randomized trial results of quality of life comparing whole abdominal irradiation and combination chemotherapy in advanced endometrial carcinoma: A gynecologic oncology group study. Qual Life Res. 2007 Feb;16(1):89-100. doi: 10.1007/s11136-006-9003-5. Epub 2006 Oct 11. PMID 17033909
- [Result] Randall ME, Filiaci VL, Muss H, Spirtos NM, Mannel RS, Fowler J, Thigpen JT, Benda JA; Gynecologic Oncology Group Study. Randomized phase III trial of whole-abdominal irradiation versus doxorubicin and cisplatin chemotherapy in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2006 Jan 1;24(1):36-44. doi: 10.1200/JCO.2004.00.7617. Epub 2005 Dec 5. PMID 16330675
- [Result] Randall ME, Brunetto G, Muss H, et al.: Whole abdominal radiotherapy versus combination doxorubicin-cisplatin chemotherapy in advanced endometrial carcinoma: a randomized phase III trial of the Gynecologic Oncology Group. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-3, 2, 2003.
- [Result] Waltkins-Bruner D, Barsevick A, Tian C, et al.: Quality of life trade-off to incremental gain in survival on Gynecologic Oncology Group (GOG) Protocol 122: whole abdominal irradiation (WAI) vs. doxorubicin-platinum (AP) chemotherapy in advanced endometrial cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1803, 449, 2003.